CLINICAL TRIAL: NCT03511079
Title: Impact of Perioperative Music on Quality of Life Measures and Biomarker Levels in Breast Cancer Patients
Brief Title: Music as a Perioperative Therapy in Breast Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruiting due to staffing and Covid-19
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kristine Widders, Assistant Professor of Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007842
Record Dates: First submitted 2018-03-14; First posted 2018-04-27 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: Music
MeSH Terms: conditions — Breast Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: There will be two groups. The intervention group will listen to music each night several days before and after surgery. The control group will not listen to music each night around the time of surgery.
Masking Description: There will be no blinding in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): This group will be given a subscription to Pandora Plus for the duration of the study. Beginning two nights before surgery, they will listen to a music playlist they created for 30 minutes prior to going to sleep. This will continue each night with the final time being 6 nights after surgery.
  Interventions: Behavioral: Music
- Control (No Intervention): This group will not listen to music each night for the duration of the study.

INTERVENTIONS:
Behavioral: Music — Music will be delivered through Pandora Plus radio via patient's computer or smartphone. The patient will choose a favorite song to create a playlist which will be used for the duration of the entire study. The subgenre of the initial song will be recorded.
  Other Names: Pandora Plus
  Arms: Music

SUMMARY:
Music has often been used in hospitals as a therapy but there is a limited amount of research looking at how music actually affects the different molecules in the body, such as cortisol (a marker of stress). There is especially a lack of research in the context of surgery. The hope is that this study will show that music can be used to minimize some of the side effects related to breast surgery and improve the patient experience.

DETAILED DESCRIPTION:
In medical practice, an ideal therapy should have maximal benefit with minimal risk. While considerable effort is being placed into discovering more effective pharmaceuticals, there is a growing field of interest in alternative therapies. In the 1970's, George Engle put forward the idea of the biopsychosocial response in which the patient's social and psychological factors can influence the body's biologic function and vice versa. One such potential therapy that could work by this mechanism is music. Advantages of music include low cost, availability, no required expertise, and minimal side effects. Studies have shown that music leads to reduced postoperative pain, anxiety, and analgesic needs in surgical patients. It has also been shown that patient selected music has greater outcomes than researcher selected music. While there is a significant body of literature on changes in clinical measurements, there are only two studies known to us which try to examine the effects of music on a molecular level, measuring cortisol and blood glucose respectively. Neither of these studies have been performed in patients undergoing surgery for breast cancer.

On the other hand, considerable research is currently being conducted to determine biomarkers in the context of surgery that are associated with poor outcomes, especially in the context of breast surgery. Stress, usually associated with cortisol levels, has been associated with increased sleep disruption, increased metabolism, increased risk of thromboembolic events, and impaired wound healing in patients. In breast cancer patients, it has been found that C-reactive protein levels correlated in fatigue postoperatively and decreased diurnal variation in cortisol has been associated with depression. Melatonin, in general, is a marker for circadian rhythm and would also be representative of sleep disruption. C-reactive protein is primarily a marker of inflammation which in turn is associated with disease progression and poorer clinical outcomes in breast surgery patients.

This study aims to determine both if music affects molecular mechanisms through measurement of clinical biomarkers as well as if there is an association with significant quality of life measures. A positive association could provide evidence into music being used as an adjunct therapy peri-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage 0 to stage III breast cancer as classified by the American Joint Committee on Cancer
* Undergoing a mastectomy or lumpectomy at Penn State Hershey Medical Center
* Fluent in written and spoken English

Exclusion Criteria:

* Hearing loss or other difficulties hearing that, in the opinion of the research team, prevent the subject from listening to music
* Serious oral health or dental conditions that affect saliva production
* Patients who have undergone pre-operative chemotherapy or pre-operative radiation therapy
* Should not be taking supplements of melatonin or taking corticosteroids
* History of liver cancer
* History of liver disease or cirrhosis (based on MELD score)
* History of endocrine tumors
* Lack of electronic device (smartphone, computer, etc) on which to listen to music
* Cognitive impairment
* Prisoner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Change in Pain | The survey will be given three days prior to surgery and seven days after surgery.
  Pain will be measured using select questions from the BREAST-Q model. The individual pain items will be measured on a 5 point Likert scale as follows:
  1. = None of the time
  2. = A little of the time
  3. = Some of the time
  4. = Most of the time
  5. = All of the time
  Total summed scores range from 12 to 60 in breast conserving modules and 16 to 80 for mastectomy modules. Higher scores are representative of more pain experienced by the patient.
Change in Sleep Quality | The scale will given three days prior to surgery and seven days after surgery.
  Sleep quality will be measured by the Karolinska Sleepiness scale. The KSS is a 9-point Likert scale often used when conducting studies involving self-reported, subjective assessment of an individual's level of drowsiness at the time. The KSS Scores are defined as follows:
  9. Extremely sleepy, fighting sleep 8. Sleepy, some effort to keep alert 7. Sleepy, but no difficulty remaining awake 6. Some signs of sleepiness 5. Neither alert nor sleepy 4. Rather alert 3. Alert 2. Very alert
  1. Extremely alert
  Higher values indicate a higher level of drowsiness.
Change in Depression | The questionnaire will be given three days prior to surgery and seven days after surgery.
  Depression will be measured with the Center for Epidemiologic Studies-Depression scale. The CES-D scale is a 20-item measure that measures how often over the past week one has experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely.
  Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Total summed scores range from 0 to 60, with high scores indicating greater depressive symptoms.

SECONDARY OUTCOMES:
Change in Salivary Cortisol level | Samples will be taken two days before surgery (AM and PM), the day of surgery (AM only), one day after surgery (AM and PM), and seven days after surgery (AM and PM).
  Samples will be taken 30 minutes after awakening (AM) and 30 minutes prior to falling asleep (PM) on select days (except the evening of the day of surgery).
Change in Salivary Melatonin level | Samples will be taken two days before surgery (AM and PM), the day of surgery (AM only), one day after surgery (AM and PM), and seven days after surgery (AM and PM).
  Samples will be taken 30 minutes after awakening (AM) and 30 minutes prior to falling asleep (PM) on select days (except the evening of the day of surgery).
Change in Salivary C-reactive protein level | Samples will be taken two days before surgery (AM and PM), the day of surgery (AM only), one day after surgery (AM and PM), and seven days after surgery (AM and PM).
  Samples will be taken 30 minutes after awakening (AM) and 30 minutes prior to falling asleep (PM) on select days (except the evening of the day of surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Kristine L Widders, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Breast Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borrell-Carrio F, Suchman AL, Epstein RM. The biopsychosocial model 25 years later: principles, practice, and scientific inquiry. Ann Fam Med. 2004 Nov-Dec;2(6):576-82. doi: 10.1370/afm.245. PMID 15576544
- [Background] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Nilsson U, Unosson M, Rawal N. Stress reduction and analgesia in patients exposed to calming music postoperatively: a randomized controlled trial. Eur J Anaesthesiol. 2005 Feb;22(2):96-102. doi: 10.1017/s0265021505000189. PMID 15816586
- [Background] Vetter D, Barth J, Uyulmaz S, Uyulmaz S, Vonlanthen R, Belli G, Montorsi M, Bismuth H, Witt CM, Clavien PA. Effects of Art on Surgical Patients: A Systematic Review and Meta-analysis. Ann Surg. 2015 Nov;262(5):704-13. doi: 10.1097/SLA.0000000000001480. PMID 26583656
- [Background] Orre IJ, Reinertsen KV, Aukrust P, Dahl AA, Fossa SD, Ueland T, Murison R. Higher levels of fatigue are associated with higher CRP levels in disease-free breast cancer survivors. J Psychosom Res. 2011 Sep;71(3):136-41. doi: 10.1016/j.jpsychores.2011.04.003. Epub 2011 May 18. PMID 21843747
- [Background] Bouchard LC, Antoni MH, Blomberg BB, Stagl JM, Gudenkauf LM, Jutagir DR, Diaz A, Lechner S, Gluck S, Derhagopian RP, Carver CS. Postsurgical Depressive Symptoms and Proinflammatory Cytokine Elevations in Women Undergoing Primary Treatment for Breast Cancer. Psychosom Med. 2016 Jan;78(1):26-37. doi: 10.1097/PSY.0000000000000261. PMID 26569533
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922